CLINICAL TRIAL: NCT05407714
Title: A Real Word Study to Evaluate the Safety and Performance of SpaceOAR System When Used to Create Space Between the Rectum and Prostate in Men Undergoing Radiotherapy for Localized T1-T2 Prostate Cancer in China
Brief Title: SpaceOAR System RWS in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0720
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Localized T1-T2 Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SpaceOAR Treatment Arm (Experimental): Single arm, up to 20 subjects with a pathologically confirmed diagnosis of clinical stage T1 or T2 prostate cancer indicated for radiotherapy will be enrolled, for there are chances of missing data in the real world study. A sample of 14 subjects provides at least 90% power for the primary objective.
  Interventions: Device: SpaceOAR Treatment

INTERVENTIONS:
Device: SpaceOAR Treatment — SpaceOAR System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of SpaceOAR System to reduce the radiation dose delivered to the anterior rectum.
  The SpaceOAR System is composed of biodegradable material and maintains space for the entire course of prostate radiotherapy treatment and is completely absorbed by the patient's body over time.

SUMMARY:
This study aims to evaluate the safety and performance of SpaceOAR System when it is used to create space between the rectum and prostate in men undergoing radiotherapy for localized T1-T2 prostate cancer in China via collecting the real word data of SpaceOAR System used, to generate local clinical evidence on Chinese patients.

DETAILED DESCRIPTION:
This study is a retrospective and prospective, single arm, real world study. For those patients who have already received the SpaceOAR treatment before study kick-off, the data at baseline and the day of procedure will be retrospectively collected. For those patients who will receive SpaceOAR treatment after study kick-off, the clinical data at baseline, the day of procedure and 30 days post procedure will be prospectively collected.

Up to 20 subjects with a pathologically confirmed diagnosis of clinical stage T1 or T2 prostate cancer indicated for radiotherapy will be enrolled, for there are chances of missing data in the real world study. A sample of 14 subjects provides at least 90% power for the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Subjects has provided the written informed consent, willing to participate in clinical data collection and willing to receive visit at 30 days post procedure. (for subjects enrolled prospectively)
* Subjects must have been pathologically confirmed prostate cancer with clinical stage T1-T2, and have been treated or will be treated with Space OAR Hydrogel in hospital in Hainan Boao Lecheng medical pilot zone.

Exclusion Criteria- no specific exclusion criteria unless the patients refuse to sign the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujun Han, Principal Investigator — Boao Yiling Life Care Center
Locations (1):
- Boao First Life Care Center-Hospital, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled 15 subjects, and collected 14 cases valid data .
Groups:
- SpaceOAR Treatment Arm: Single arm, up to 20 subjects with a pathologically confirmed diagnosis of clinical stage T1 or T2 prostate cancer indicated for radiotherapy will be enrolled, for there are chances of missing data in the real world study. A sample of 14 subjects provides at least 90% power for the primary objective.
  SpaceOAR Treatment: SpaceOAR System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of SpaceOAR System to reduce the radiation dose delivered to the anterior rectum.
  The SpaceOAR System is composed of biodegradable material and maintains space for the entire course of prostate radiotherapy treatment and is completely absorbed by the patient's body over time.
Period: Overall Study
Arm/Group | SpaceOAR Treatment Arm
Started | 15
Cases of Valid Data | 14
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SpaceOAR Treatment Arm
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 15

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: The distance between the posterior prostatic capsule and anterior rectal wall,
Time Frame: Within 10 days post spaceOAR hydrogel administration.
Population: The distance between the posterior prostatic capsule and anterior rectal wall is measured on the axial image slice closest to halfway between apex and base, from posterior edge of prostate to inner rectal wall via MRI.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SpaceOAR Treatment Arm
Number analyzed (Participants) | 14
mm | 15.1 (1.8)

2. Primary Outcome: Primary Safety Endpoint
Description: Subjects with AEs related to SpaceOAR system and/or procedure within 30 days following procedure will be observed.
Time Frame: Within 30 days following procedure
Measure: Count of Participants; unit: Participants
Groups:
- SpaceOAR Treatment Arm: Enrolled 15 subjects
Arm/Group | SpaceOAR Treatment Arm
Number analyzed (Participants) | 15
Participants | 2

3. Secondary Outcome: Functional Success
Description: Distance Posterior Prostatic Capsule and Anterior Rectal Wall
Time Frame: Within 10 days post spaceOAR hydrogel administration.
Population: Creation of at least 7.5mm space between the posterior prostatic capsule and anterior rectum wall via comparative pre and post SpaceOAR hydrogel injection MRI scans.
Measure: Count of Participants; unit: Participants
Arm/Group | SpaceOAR Treatment Arm
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Time Frame: 30 days post procedure.
Arm/Group | SpaceOAR Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SpaceOAR Treatment Arm (N=15)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT05407714/Prot_004.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT05407714/SAP_005.pdf